CLINICAL TRIAL: NCT01042899
Title: Rehabilitation Research and Training Center for Traumatic Brain Injury Interventions
Brief Title: Rehabilitation Research and Training Center for Traumatic Brain Injury Interventions--Teen Online Problem Solving Study
Acronym: RRTC--TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: MetroHealth Medical Center (Other); Nationwide Children's Hospital (Other); Rainbow Babies and Children's Hospital (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H133B090010--01
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; intracranial edema; brain edema; craniocerebral trauma; head injury; brain hemorrhage, traumatic; subdural hematoma; brain concussion; head injuries, closed; epidural hematoma; extra-axial hemorrhage; cortical contusion; wounds and injuries; disorders of environmental origin; trauma, nervous system; brain injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Craniocerebral Trauma; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Brain Concussion; Head Injuries, Closed; Hematoma, Epidural, Spinal; Brain Contusion; Wounds and Injuries; Disorders of Environmental Origin; Trauma, Nervous System; Brain Injuries | interventions — TOPS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Teen Online Problem Solving (TOPS) (Experimental): Web intervention
  Interventions: Behavioral: Teen Online Problem Solving (TOPS); Behavioral: Teen Online Problem Solving--Teen Only (TOPS-TO); Behavioral: Internet Resources Comparison (IRC)
- Teen Online Problem Solving---Teen Only (Experimental): Web Intervention
  Interventions: Behavioral: Teen Online Problem Solving--Teen Only (TOPS-TO)
- Internet Resources Comparison (Active Comparator): Web Intervention
  Interventions: Behavioral: Internet Resources Comparison (IRC)

INTERVENTIONS:
Behavioral: Teen Online Problem Solving (TOPS) — The TOPS program has 10 sessions that provide training in stress management, problem solving, communication, and social skills to all enrolled families, while the remaining 6 sessions address content related to the stressors and burdens of individual families. Each self-guided online session includes real adolescents talking about how TBI affected them, content regarding the skill, video clips showing adolescents and/or families modeling the skill, and exercises giving the family an opportunity to practice the skill. After the completion of the self-guided web pages, the family will meet with the therapist via videoconference; the therapist will review the exercises and help the family implement the problem-solving process with a problem or goal identified by the family.
  Other Names: TOPS
  Arms: Teen Online Problem Solving (TOPS)
Behavioral: Teen Online Problem Solving--Teen Only (TOPS-TO) — TOPS-TO targets the same skills as TOPS and includes largely the same website and intervention content. However, it differs with respect to the extent of family involvement in the sessions. In TOPS-TO, sessions will be conducted with the child or adolescent alone, rather than with the family as whole. Parents will be given access to the TOPS-TO website content via their own password protected site so they will understand the skills that their child is learning. However, only the adolescent, and not the parents, will participate in the synchronous videoconferences with the therapist.
  Other Names: TOPS-TO
  Arms: Teen Online Problem Solving (TOPS); Teen Online Problem Solving---Teen Only
Behavioral: Internet Resources Comparison (IRC) — Families in the IRC group will also receive a computer, printer, and high-speed internet access if they do not currently have these. Additionally, IRC families receive access to a home page of brain injury resources and links (identical to those given on the TOPS and TOPS-TO homepage) but will not be able to access specific session content. This will enable us to equate the groups with respect to access to the information and resources available on the Web.
  Other Names: IRC
  Arms: Internet Resources Comparison; Teen Online Problem Solving (TOPS)

SUMMARY:
This study will evaluate the effectiveness of an Internet-based psychosocial treatment in improving problem-solving, communication skills, stress management strategies, and coping among teens who have had a traumatic brain injury and their families.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) in adolescents is a significant stressor for both the teen and his or her family. Existing interventions are rare and access to treatment can be restricted by distance and finances. Based on previous findings and participant feedback, we propose to expand the previously developed TOPS intervention by conducting a multi-site study comparing the efficacy of TOPS to that of TOPS-Teen Only (TOPS-TO) in improving child behavior and functioning, parental depression and distress and family functioning. The efficacy of both active treatments would be examined in relation to an internet resource comparison group (IRC). During years 1-3, we will recruit 165 children between the ages of 11 and 18 with moderate to severe TBI and randomly assign them to receive TOPS, TOPS-TO, or IRC. We anticipate that TOPS will result in improvements in child, caregiver, and family functioning relative to IRC; but that TOPS-TO will only result in improvements in child behavior and adjustment. Based on prior research, we anticipate that the family-level treatment model of TOPS may be more effective than TOPS-TO in improving child behavior for children/adolescents with fewer social resources. Given these expectations, we will test the following hypotheses: 1) Children with TBI receiving either TOPS or TOPS-TO will have fewer behavior problems, greater social competence, and better functioning than those receiving IRC at both post-treatment and at a 6-month follow-up assessment. 2) Caregivers of children receiving TOPS will report less depression and psychological distress, less parent-child conflict, and better family functioning than those receiving TOPS-TO or IRC at both post-treatment and at a 6-month follow-up assessment. 3) Social resources will moderate treatment efficacy, such that children with limited social and economic resources will show greater improvements in the more comprehensive TOPS intervention. We hypothesize better teen problem solving and communication skills, fewer teen emotional/behavioral problems, less parental burden and distress, and less parent-teen conflict at follow-up among the TOPS group compared to the IRC group. TOPS makes use of emerging technology to address the multifaceted needs of teens following TBI with the goal of improving the teen's social and emotional functioning, thereby enabling him or her to better negotiate the complex transition to adulthood and independent functioning.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe TBI that occurred within the last 18 months
* Overnight hospital stay
* English-speaking
* Parent must be willing to provide informed consent

Exclusion Criteria:

* Child does not live with parents or guardian
* Child or parent has history of hospitalization for psychiatric problem
* TBI is a result of child abuse
* Child suffered a non-blunt injury (e.g., projectile wound, stroke, drowning, or other form of asphyxiation)
* Diagnosed with moderate or severe mental retardation, autism, or a significant developmental disability

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2010-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Parent Report Measures | 5 years

SECONDARY OUTCOMES:
Teen Self-Report Measures | 5 years
Neuropsychological Testing | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharil L Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - The Children's Hospital, Denver, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies' and Children's Hospital, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Narad ME, Kaizar EE, Zhang N, Taylor HG, Yeates KO, Kurowski BG, Wade SL. The Impact of Preinjury and Secondary Attention-Deficit/Hyperactivity Disorder on Outcomes After Pediatric Traumatic Brain Injury. J Dev Behav Pediatr. 2022 Aug 1;43(6):e361-e369. doi: 10.1097/DBP.0000000000001067. Epub 2022 Feb 15. PMID 35170571
- [Derived] Wade SL, Fisher AP, Kaizar EE, Yeates KO, Taylor HG, Zhang N. Recovery Trajectories of Child and Family Outcomes Following Online Family Problem-Solving Therapy for Children and Adolescents after Traumatic Brain Injury. J Int Neuropsychol Soc. 2019 Oct;25(9):941-949. doi: 10.1017/S1355617719000778. Epub 2019 Aug 13. PMID 31405391
- [Derived] Narad ME, Raj S, Yeates KO, Taylor HG, Kirkwood MW, Stancin T, Wade SL. Randomized Controlled Trial of an Online Problem-Solving Intervention Following Adolescent Traumatic Brain Injury: Family Outcomes. Arch Phys Med Rehabil. 2019 May;100(5):811-820. doi: 10.1016/j.apmr.2019.01.010. Epub 2019 Feb 6. PMID 30738021
- [Derived] Wade SL, Kaizar EE, Narad M, Zang H, Kurowski BG, Yeates KO, Taylor HG, Zhang N. Online Family Problem-solving Treatment for Pediatric Traumatic Brain Injury. Pediatrics. 2018 Dec;142(6):e20180422. doi: 10.1542/peds.2018-0422. Epub 2018 Nov 9. PMID 30413559
- [Derived] Lantagne A, Peterson RL, Kirkwood MW, Taylor HG, Stancin T, Yeates KO, Wade SL. Featured Article: Interpersonal Stressors and Resources as Predictors of Adolescent Adjustment Following Traumatic Brain Injury. J Pediatr Psychol. 2018 Aug 1;43(7):703-712. doi: 10.1093/jpepsy/jsy020. PMID 29617953
- [Derived] Wade SL, Narad ME, Kingery KM, Taylor HG, Stancin T, Kirkwood MW, Yeates KO. Teen online problem solving for teens with traumatic brain injury: Rationale, methods, and preliminary feasibility of a teen only intervention. Rehabil Psychol. 2017 Aug;62(3):290-299. doi: 10.1037/rep0000160. PMID 28836809
- [Derived] Wade SL, Cassedy AE, Fulks LE, Taylor HG, Stancin T, Kirkwood MW, Yeates KO, Kurowski BG. Problem-Solving After Traumatic Brain Injury in Adolescence: Associations With Functional Outcomes. Arch Phys Med Rehabil. 2017 Aug;98(8):1614-1621. doi: 10.1016/j.apmr.2017.03.006. Epub 2017 Apr 4. PMID 28389109